CLINICAL TRIAL: NCT01217372
Title: A Prospective, Randomized, Open Blind Endpoint (Probe) Trial to Assess the Possibility to Prevent Stone Recurrence by Lemon Juice Supplementation in Patients With Recurrent Calcium Oxalate Nephrolithiasis (LIMONE Study)
Brief Title: Nephrolithiasis Prevention by Lemon Juice
Acronym: LIMONE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LIMONE
Record Dates: First submitted 2010-09-30; First posted 2010-10-08 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Nephrolithiasis
Keywords: Recurrent idiopathic calcium oxalate nephrolithiasis.
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lemon supplementation YES (Experimental): 60 ml of lemon juice twice daily (an amount expected to provide 6 grams or 92 mEq of citric acid per day)
  Interventions: Dietary Supplement: Lemon supplementation
- Lemon supplementation NO (No Intervention): No lemon supplementation

INTERVENTIONS:
Dietary Supplement: Lemon supplementation — 60 ml of lemon juice twice daily (an amount expected to provide 6 grams or 92 mEq of citric acid per day)
  Arms: Lemon supplementation YES

SUMMARY:
Calcium oxalate nephrolithiasis is a relatively common disease. The prevalence in the general population may range from 10 to 12 percent, and 0.4 to 1 percent of new cases are reported every year according to different series. Without specific pharmacological therapy, the recurrence rate in patient with established diagnosis of nephrolithiasis is extremely high and may range from 15 to 20 percent per year, with a cumulative incidence at five years ranging from 27 to 50 percent.Although genetic factors play an important role in the development of nephrolithiasis, environmental factors such as diet also appear to affect stone formation. Potassium citrate is also effective in preventing stone recurrence in patients with calcium oxalate nephrolithiasis. Low tolerability, however, may remarkably limit the use of these medication. Citrus fruits are a natural rich source of citrate and diet supplementation with juice of citrus fruits may represent a valuable alternative option to supply citrate without exposing the patients to the adverse effects of citrate containing medications. Among the most commonly consumed citrus fruits, lemons contain the greatest concentrations of citric acid (49,2 g/Kg);a half cup of pure lemon juice can provide a daily amount of citrate comparable to that of a standard daily dose of alkali citrate medications.

A few studies tried to evaluate the effects of lemon juice supplementation in patients with calcium oxalate nephrolithiasis, but the findings were flawed by the retrospective, observational design of the study or by the too small sample size that limited the power of statistical analyses and the reliability of the results. This study will be primarily aimed at evaluating whether lemon juice added to standard diet recommendations compared to diet recommendations alone may reduce the risk of new stone formation in patients with recurrent idiopathic calcium oxalate nephrolithiasis. Secondarily, the study will evaluate the effects of lemon juice supplementation on complications of nephrolithiasis such as urinary tract infections, colic symptoms, and hospitalizations for stone disruption or removal, as well as the effects on urinary factors (such as urinary citrate, oxalate, calcium excretion or pH) that may favor or limit stone formations and the relationships between these effects and the risk of stone recurrence.

DETAILED DESCRIPTION:
BACKGROUND Calcium oxalate nephrolithiasis is a relatively common disease. The prevalence in the general population may range from 10 to 12 percent, and 0.4 to 1 percent of new cases are reported every year according to different series. Without specific pharmacological therapy, the recurrence rate in patient with established diagnosis of nephrolithiasis is extremely high and may range from 15 to 20 percent per year, with a cumulative incidence at five years ranging from 27 to 50 percent.

Although genetic factors play an important role in the development of nephrolithiasis, environmental factors such as diet also appear to affect stone formation. Diet based on restricted intake of animal proteins and salt, combined with a normal calcium intake, may reduce the risk of stone formation. However, the efficacy in preventing stone recurrences is limited, in particular in repeated stone formers.

Potassium citrate is also effective in preventing stone recurrence in patients with calcium oxalate nephrolithiasis. Low tolerability, however, may remarkably limit the use of these medication.

Citrus fruits are a natural rich source of citrate and diet supplementation with juice of citrus fruits may represent a valuable alternative option to supply citrate without exposing the patients to the adverse effects of citrate containing medications.

Among the most commonly consumed citrus fruits, lemons contain the greatest concentrations of citric acid (49,2 g/Kg), nearly 5 times the concentrations in the orange. A half cup of pure lemon juice can provide a daily amount of citrate comparable to that of a standard daily dose of alkali citrate medications. The citrate supplied with the juice that escapes metabolic degradation in vivo is excreted unchanged in the urine where may prevent the tendency of calcium oxalate salts to precipitate. Lemon juice supplementation may also have the additional advantage of reducing urinary calcium excretion without affecting oxalate excretion, while orange juice does not affect urinary calcium and may increase urinary oxalate.

A few studies tried to evaluate the effects of lemon juice supplementation in patients with calcium oxalate nephrolithiasis, but the findings were flawed by the retrospective, observational design of the study or by the too small sample size that limited the power of statistical analyses and the reliability of the results. Thus, the protective effect of lemon juice supplementation against recurrence of stones in patients with calcium oxalate nephrolithiasis is worth investigating in adequately powered and designed trials.

AIM The study will be primarily aimed at evaluating whether lemon juice added to standard diet recommendations compared to diet recommendations alone may reduce the risk of new stone formation in patients with recurrent idiopathic calcium oxalate nephrolithiasis. Secondarily, the study will evaluate the effects of lemon juice supplementation on complications of nephrolithiasis such as urinary tract infections, colic symptoms, and hospitalizations for stone disruption or removal, as well as the effects on urinary factors (such as urinary citrate, oxalate, calcium excretion or pH) that may favor or limit stone formations and the relationships between these effects and the risk of stone recurrence.

DESIGN

According to urinary citrate excretion at baseline evaluation patients satisfying the selection criteria will be stratified into two strata:

Stratum 1: Hypocitraturia (urinary citrate excretion >320 mg/24 h) Stratum 2: Normocitraturia (urinary citrate excretion <320 mg/24 h) Within each stratum, patients will be randomized on a 1:1 basis to two-year treatment with lemon juice supplemented to standard recommended diet or to standard diet alone. All patients in the hypocitraturic stratum will also be prescribed potassium citrate 2g twice daily. Due to the Prospective, Randomized, Open, Blind Endpoint (PROBE) design of the study, patients and physicians in charge of patient care and monitoring will be aware of patient treatment, while all the Investigators involved in data handling and analyses will be blinded to patient treatment allocation.

101 patients per group will have to be included. Thus, a total of 202 patients will have to be randomized.

ELIGIBILITY:
Inclusion Criteria:

* male and female >18 years
* history of recurrent nephrolithiasis, with one o more calcium oxalate or mixed (calcium oxalate and phosphate, calcium oxalate and uric acid) stone formation over the last 5 years
* at least one kidney stone at baseline documented by renal echography and/or X-ray evaluation.
* written informed consent

Exclusion Criteria:

* Obstructive uropathy, chronic urosepsis, renal failure (serum creatinine >1.8 mg/dl), renal tubular acidosis, primary hyperparathyroidism, primary hyperoxaluria, pure uric acid and cystine stones, medullary sponge kidney
* lithotripsy treatment within the last 6 months
* active peptic ulcer disease, gastric esophagus reflux
* concomitant clinical conditions that might affect completion of the study or jeopardize data interpretation
* pharmacological therapy for stone disease over the last month
* impossibility to assess the number of kidney stones
* inability to provide an informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
Spontaneous passage of stone or gravel. | At 6 month.
Appearance of new stones. | At 6 month.
More than 30 percent increase in pre-existing stone size | At 6 month.
Spontaneous passage of stone or gravel. | At 12 month.
Spontaneous passage of stone or gravel. | At 24 month.
Appearance of new stones. | At 12 month.
Appearance of new stones. | At 24 month.
More than 30 percent increase in pre-existing stone size | At 12 month.
More than 30 percent increase in pre-existing stone size | At 24 month.

CONTACTS AND LOCATIONS:
Locations (1):
- Unit of Nephrology and Dialysis, Bergamo, Italy